CLINICAL TRIAL: NCT05697783
Title: Methadone vs. Transdermal Fentanyl for Opioid Withdrawal Syndrome : Comparison of Two Groups of Intubated and Ventilated Patients in the Intensive Care Unit: Before-after Intervention Study
Brief Title: Methadone vs. Transdermal Fentanyl for Opioid Withdrawal Syndrome
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, sara dichtwald, Dr, Meir Medical Center
Other Study IDs: 0008-23-MMC
Record Dates: First submitted 2023-01-04; First posted 2023-01-26 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Delirium in the Intensive Care Unit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Methadone-treated group
  Interventions: Drug: Administration of methadone instead of fentanyl patch
- Fentanyl-patch treated group

INTERVENTIONS:
Drug: Administration of methadone instead of fentanyl patch — comparison of delirium rates in methadone vs fentanyl patch treated patients
  Other Names: comparison of delirium rates in methadone vs fentanyl patch treated patients
  Groups: Methadone-treated group

SUMMARY:
Many patients in the general intensive care unit experience pain, as a result of an injury or underlying disease, surgery or an invasive procedure.

Pain management is an integral part of the treatment of critical patients, and this is first and foremost to alleviate their suffering. Along with this, there is another therapeutic benefit in the form of relief from symptoms accompanying pain such as an increase in oxygen consumption, immune changes, hyper metabolism etc.

Currently, the pain treatment is based on a multi-modal analgesia approach in which drugs from several drug groups and different mechanisms are given, in order to relieve the pain by suppressing several nerve and inflammatory pathways. However, the treatment is still based on opioids, despite multiple adverse effects, including tolerance and withdrawal syndrome.

Opioids affect several receptors, mainly the µ receptor, in an agonistic, antagonistic or agonistic-antagonistic manner. The main opioids used for pain relief in the intensive care unit are morphine, fentanyl and remifentanil.

After prolonged treatment with opioids, a sudden cessation of their use will result in a withdrawal syndrome which will manifest itself in delirium, restlessness, hypertension, anxiety, sweating, vomiting etc. (2-3). In order to avoid the withdrawal syndrome, the dose must be tapered down gradually, often using alternative long-term opioids, such as methadone and buprenorphine (-4).

In the general intensive care unit at our institution, patients were treated with fentanyl patches in decreasing doses in order to lead the patient safely through the withdrawal syndrome, while trying to reduce the negative physiological effects as much as possible. In November 2021, we started using oral methadone instead of fentanyl patches, as a long acting opioid, as used in many ICU's worldwide, in order to avoid withdrawal syndrome in patients who received continuous infusion of short-acting opioids, such as remifentanil, for long periods of time while being intubated and ventilated. In the past year since the methadone treatment was started, 50 patients were treated in the unit with methadone with the indication of relieving the withdrawal symptoms from opioids.

We intent to investigate whether there is a difference in the incidence of delirium in patients who were treated with methadone vs patients who were treated with fentanyl patches in order to alleviate withdrawal symptoms.

ELIGIBILITY:
Inclusion Criteria:All patients aged 18-99 who were treated with methadone in the intensive care unit from November 2021 to November 2022, as well as all patients aged 18-99 who were admitted to the intensive care unit from November 2020 to November 2021 and were treated with a fentanyl patch as a control group.

-

Exclusion Criteria:None

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged 18-99 who were treated with methadone in the intensive care unit from November 2021 to November 2022, as well as all patients aged 18-99 who were admitted to the intensive care unit from November 2020 to November 2021 and were treated with a fentanyl patch as a control group.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Delirium | through study completion, an average of 2 years
  Delirium as estimated by RASS score

CONTACTS AND LOCATIONS:
Locations (1):
- Meir medical center Kfar Saba, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No